CLINICAL TRIAL: NCT02073448
Title: A Multicenter, Randomized, Double-blinded, Active-controlled Parallel Group Efficacy and Safety Study of GK530G Versus CD0271 0.1% Gel and CD1579 2.5% Gel in the Treatment of Acne Vulgaris.
Brief Title: Efficacy and Safety Study of GK530G Versus CD0271 0.1% Gel and CD1579 2.5% Gel in the Treatment of Acne Vulgaris.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDT.07.SPR.27123
Record Dates: First submitted 2014-02-20; First posted 2014-02-27 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide; Adapalene; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GK530G (Experimental): Fixed-dose combination gel of Adapalene and Benzoyl Peroxide
  Interventions: Drug: GK530G
- CD0271 (Active Comparator): Adapalene 01% Gel
  Interventions: Drug: CD0271
- CD1579 (Active Comparator): Benzoyl Peroxide 2.5% Gel
  Interventions: Drug: CD1579

INTERVENTIONS:
Drug: GK530G
  Other Names: Fixed-dose combination gel of Adapalene and Benzoyl Peroxide
  Arms: GK530G
Drug: CD0271
  Other Names: Adapalene 0.1% Gel
  Arms: CD0271
Drug: CD1579
  Other Names: Benzoyl Peroxide 2.5% Gel
  Arms: CD1579

SUMMARY:
This study is to demonstrate the superiority in efficacy of the GK530G (fixed combination of CD0271 0.1% and CD1579 2.5%) versus each of the monads (CD0271 0.1% and CD1579 2.5%) in the treatment of acne vulgaris for up to 12 weeks, in the Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at the age of 12 or older at the Screening visit.
* Those with clinical diagnosis of acne vulgaris with more than 20 noninflammatory lesions (open and closed comedones) and 12 to 100 (inclusive) inflammatory lesions (papules, pustules and nodules) on the face (forehead, both cheeks, nose and chin).

Exclusion Criteria:

* Those with more than two nodular acne lesions or any cysts.
* Those with the diagnosis of any acne conglobata, any acne fulminans, any chloracne, or any drug induced acne.
* Those who have clinically significant abnormal findings or conditions on skin other than acne such as atopic dermatitis, perioral dermatitis, or rosacea that potentially interfere with study assessments according to Investigator's judgment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (13):
  - Galderma investigational site, Chitose, Hokkaido
  - Galderma investigational site, Kitami, Hokkaido
  - Galderma investigational site, Sapporo, Hokkaido
  - Galderma investigational site, Kagoshima, Kagoshima-ken
  - Galderma investigational site, Yokohama, Kanagawa
  - Galderma investigational site, Kurashiki, Okayama-ken
  - Galderma investigational site, Daitō, Osaka
  - Galderma investigational site, Neyagawa, Osaka
  - Galderma investigational site, Osaka, Osaka
  - Galderma investigational site, Sakai, Osaka
  - Galderma investigational site, Saitama, Saitama
  - Galderma investigational site, Adachi City, Tokyo
  - Galderma investigational site, Setagaya City, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- CD0271: Adapalene 01% Gel
  CD0271
- GK530G: Fixed-dose combination gel of Adapalene and Benzoyl Peroxide
  GK530G
- CD1579: Benzoyl Peroxide 2.5% Gel
  CD1579
Period: Overall Study
Arm/Group | CD0271 | GK530G | CD1579
Started | 101 | 212 | 104
Completed | 99 | 200 | 99
Not Completed | 2 | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GK530G | CD0271 | CD1579 | Total
Number analyzed (Participants) | 212 | 101 | 104 | 417
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 116 | 56 | 56 | 228
  Between 18 and 65 years | 96 | 45 | 48 | 189
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.7 (6.5) | 19.6 (6.0) | 19.3 (5.4) | 19.6 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 67 | 74 | 282
  Male | 71 | 34 | 30 | 135
Region of Enrollment [Number; unit: participants]
  Japan | 212 | 101 | 104 | 417

OUTCOME MEASURES:

1. Primary Outcome: Percent Changes From Baseline in Total Lesion Counts
Time Frame: Baseline - Week12
Measure: Median (Full Range); unit: percent change
Arm/Group | CD0271 | GK530G | CD1579
Number analyzed (Participants) | 101 | 212 | 104
percent change | 68.6 [-62.4 to 97.5] | 82.7 [-15.9 to 100] | 81.6 [-31.6 to 98.6]

2. Secondary Outcome: Percent of Subjects With Adverse Events
Time Frame: up to 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | CD0271 | GK530G | CD1579
Number analyzed (Participants) | 101 | 212 | 104
percentage of participants | 27.7 | 44.8 | 37.5

3. Secondary Outcome: Local Tolerability (Erythema)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | GK530G | CD0271 | CD1579
Number analyzed (Participants) | 212 | 101 | 104
participants
  Mild | 78 | 32 | 20
  Moderate | 24 | 5 | 4
  Severe | 2 | 0 | 1

4. Secondary Outcome: Local Tolerability (Scaling)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | GK530G | CD0271 | CD1579
Number analyzed (Participants) | 212 | 101 | 104
participants
  Mild | 105 | 37 | 24
  Moderate | 33 | 9 | 3
  Severe | 1 | 1 | 0

5. Secondary Outcome: Local Tolerability (Dryness)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | GK530G | CD0271 | CD1579
Number analyzed (Participants) | 212 | 101 | 104
participants
  Mild | 113 | 44 | 29
  Moderate | 31 | 6 | 4
  Severe | 1 | 1 | 0

6. Secondary Outcome: Local Tolerability (Pruritus)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | GK530G | CD0271 | CD1579
Number analyzed (Participants) | 212 | 101 | 104
participants
  Mild | 61 | 24 | 24
  Moderate | 21 | 2 | 9
  Severe | 3 | 0 | 1

7. Secondary Outcome: Local Tolerability (Stinging/Burning)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | GK530G | CD0271 | CD1579
Number analyzed (Participants) | 212 | 101 | 104
participants
  Mild | 106 | 49 | 21
  Moderate | 76 | 11 | 9
  Severe | 7 | 2 | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | CD0271 | GK530G | CD1579
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/212 | 0/104
Other Adverse Events (participants affected / at risk) | 28/101 | 95/212 | 39/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD0271 (N=101) | GK530G (N=212) | CD1579 (N=104)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 18 (18) | 14 (15)
Pharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (5) | 3 (4)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (4) | 5 (5) | 4 (5)
Skin irritation (Skin and subcutaneous tissue disorders) | 7 (7) | 26 (27) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Skin test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Premenstrual syndrome (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis perennial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No